CLINICAL TRIAL: NCT07371013
Title: Fecal Microbiota Transplantation in Children With Autism Spectrum Disorder and Gastrointestinal Symptoms: A Pilot Study
Brief Title: Fecal Microbiota Transplantation in Children With Autism Spectrum Disorder and Gastrointestinal Symptoms
Acronym: FMT-ASD-GI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Mother and Child, Warsaw, Poland (Other)
Collaborators: Human Biome Institute S.A. (Industry)
Responsible Party: Principal Investigator, dr n.med. Anna Liber, Head of the Department of Nutrition, Institute of Mother and Child, Warsaw, Poland
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 12/2025
Record Dates: First submitted 2026-01-12; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2025-12

CONDITIONS: Autism Spectrum Disorder; Gastrointestinal Symptoms
Keywords: fmt; asd; gi; autism
MeSH Terms: conditions — Autism Spectrum Disorder; Child Development Disorders, Pervasive; Autistic Disorder

STUDY DESIGN:
Intervention Model Description: Randomised, placebo-controlled, pilot study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MBiotix® HBI Caps (Experimental)
  Interventions: Other: MBiotix® HBI Caps
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Other: MBiotix® HBI Caps — MBiotix HBI Caps (Human Biome Institute, Poland) are enteric-coated capsules containing a concentrated suspension of gut microbiota obtained by centrifugation of a solution prepared from 60 g of donor stool suspended in 200 ml of 0.9% NaCl and glycerol. Each capsule set contains approximately 10¹³ viable bacterial cells.
  Dosing depends on body weight:
  Children weighing **>35 kg** will receive 60 g at visit 1 and 30 g at visits 2 (after 4 weeks) and 3 (after 8 weeks).
  Children weighing **<35 kg** will receive 30 g at visit 1 and 15 g at visits 2 (after 4 weeks) and 3 (after 8 weeks).
  Arms: MBiotix® HBI Caps
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The aim of the study is to evaluate the effectiveness and safety of fecal microbiota transplantation (FMT) in reducing gastrointestinal (GI) and behavioral symptoms in children with autism spectrum disorder (ASD).

Children with ASD often experience GI problems such as constipation, diarrhea, and abdominal pain. These symptoms can negatively affect their daily life and behavior. Recent research suggests that the gut microbiota-the community of bacteria and other microorganisms living in the intestines-plays an important role in digestion, immunity, and communication with the brain through the gut-brain axis. Modifying the gut microbiota may help improve GI symptoms and possibly behavioral functioning.

FMT involves giving a preparation containing gut microbiota from a healthy donor after bowel cleansing. The product used in this study is MBiotix HBI Caps, produced by Human Biome Institute. A placebo (inactive substance) will also be used for comparison. Both will be given as frozen oral capsules that look identical.

20 children aged 6-12 years will take part. Participants will be randomly assigned to receive either the microbiota preparation or placebo. The study includes several visits over about 6 months. Before the first dose, every child will undergo bowel cleansing with a special preparation (Polyethylene Glycol, PEG). During the study, participants will be asked to keep a symptom diary, complete questionnaires, and record child's diet. Biological samples (stool, urine, saliva) will be collected at specific time points for analysis. Every child will also be assessed by a psychologist before the study begins and again during the study using standardized tools (Autism Diagnostic Observation Schedule, Second Edition, ADOS-2) to evaluate behavioral functioning and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Providing informed consent for participation in the study by the child's legal representative - parent or legal guardian.
* Diagnosis of autism spectrum disorder according to DSM-5 or ICD-11 criteria.
* Ability to swallow an empty test capsule identical in shape and size to the investigational product
* Abnormal stool consistency observed by parents for at least 2 months prior to study inclusion.

Patients with an average stool consistency greater than 5 on the Bristol Stool Form Scale (BSFS) during the baseline period will be classified as having diarrhea.

Patients with an average stool consistency less than 3 on the Bristol Stool Form Scale during the baseline period will be classified as having constipation.

Exclusion Criteria:

* Presence of a gastrointestinal disease such as celiac disease, food allergy, inflammatory bowel disease, pancreatitis, chronic liver disease, eosinophilic esophagitis, peptic ulcer disease of the stomach or duodenum, Hirschsprung's disease.
* Primary or secondary immunodeficiency, including absolute neutrophil count in peripheral blood <1500 measured within 28 days prior to planned FMT.
* History of surgery involving disruption of intestinal continuity within 3 months prior to study inclusion.
* Lactose or fructose intolerance. Patients with lactose intolerance who follow an elimination diet and still experience symptoms may be included in the study.
* Malnutrition defined as Body Mass Index (BMI) below the 3rd percentile based on Polish growth charts from 2010.
* Overweight or obesity defined as BMI above the 85th percentile based on Polish growth charts from 2010.
* Active infection requiring antibiotic therapy.
* Expected use of antibiotics during participation in the study.
* Use of probiotics during participation in the study.
* Inability to undergo bowel cleansing therapy (Dicopeg Endo).
* Inability to swallow an empty test capsule.
* Lack of consent from the child's legal representative - parent or legal guardian - for participation in the study.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Number of patients who showed an improvement in stool consistency by at least 1 point on the Bristol Stool Scale compared to the baseline period. | 4,8,9,12,26,20 weeks
  The average stool consistency will be calculated from the one-week baseline period and from weekly observation periods during the study.

SECONDARY OUTCOMES:
Bowel movements | 4,8,9,12,16,20 weeks
  Change in the number of bowel movements compared to the baseline period.
Abdominal pain episodes | 4,8,9,12,16,20 weeks
  Change in the number of abdominal pain episodes compared to the baseline period.
Days with abdominal pain | 4,8,9,12,16,20 weeks
  Change in the number of days with abdominal pain compared to the baseline period. Endpoints assessing abdominal pain will be evaluated only in children who are able to communicate their symptoms.
Excessive gas | 4,8,9,12,16,20 weeks
  Change in the number of days with excessive gas according to parent's assessment.
Regurgitation | 4,8,9,12,16,20 weeks
  Change in the number of days with regurgitation compared to the baseline period.
Vomiting | 4,8,9,12,16,20 weeks
  Change in the number of days with vomiting compared to the baseline period.
Child absence | 4,8,9,12,16,20 weeks
  Change in the number of days absent from kindergarten or school due to symptoms.
Parent's work absence | 4,8,9,12,16,20 weeks
  Change in the number of days of parental or caregiver work absence due to symptoms
Adverse events | 0,4,8,9,12,16,20 weeks
  Adverse events reported by children and parents, recorded in the symptom diary and reported to the physician.
SRS-2 | 9,20 weeks
  Change in the score of the psychological test Social Responsiveness Scale-2 (SRS-2) compared to baseline.
ASRS | 9,20 weeks
  Change in the score of the psychological test Autism Spectrum Rating Scales (ASRS) compared to baseline
ADOS-2 | 9,20 weeks
  Change in the score of the psychological test Autism Diagnostic Observation Schedule-2 (ADOS-2) compared to baseline.
CBCL | 9,20 weeks
  Change in the score of the psychological test Child Behavior Checklist (CBCL) compared to baseline.
ABAS-3 | 9,20 weeks
  Change in the score of the psychological test Adaptive Behavior Assessment System-3 (ABAS-3) compared to baseline.
QoLA | 9,20 weeks
  Change in parental quality of life assessed using the Quality of Life in Autism Questionnaire (QoLA) compared to baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Mother and Child, Warsaw, Masovian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Yes
IPD used in the results publication